CLINICAL TRIAL: NCT05959096
Title: Effect of Injection Site on the Relative Bioavailability of a Single Dose of LY3437943 in Healthy Participants With a High Body Mass Index
Brief Title: A Study of LY3437943 in Healthy Participants With a High Body Mass Index
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18532; J1I-MC-GZBS (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Healthy
MeSH Terms: interventions — retatrutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3437943 (Part A) (Experimental): LY3437943 administered subcutaneously (SC) in either thigh, upper arm, or abdomen
  Interventions: Drug: LY3437943
- LY3437943 (Part B) (Experimental): LY3437943 administered intravenously (IV)
  Interventions: Drug: LY3437943

INTERVENTIONS:
Drug: LY3437943 — Administered SC
  Arms: LY3437943 (Part A)
Drug: LY3437943 — Administered IV
  Arms: LY3437943 (Part B)

SUMMARY:
The study is conducted in two parts (Part A and B). The main purpose of this study is to look at the amount of the LY3437943 that gets into the blood stream and how long it takes the body to get rid of it when given subcutaneously (SC, under the skin) in the upper arm and thigh compared to the abdomen in healthy participants with high body mass index (BMI) in Part A. In Part B, the participants receive LY3437943 intravenously (IV, through a vein) where the safety and tolerability of LY3437943 are evaluated and information about any side effects experienced will be collected. For each participant, the total duration of the study will be approximately up to 157 days and 99 days for Part A and Part B, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females of nonchildbearing potential as determined by medical history, physical examination, and other screening procedures
* Body mass index (BMI) between 27.0 and 45.0 kilograms per meter squared (kg/m²), inclusive
* Are agreeable to receiving study treatment by injections under the skin or through a vein.

Exclusion Criteria:

* Have a history of diabetes (except gestational diabetes) or current diagnosis of diabetes (any form)
* Have a significant history of, or presence of, any of the following disorders capable of significantly altering the absorption, metabolism, or elimination of drugs
* Have known allergies to LY3437943, related compounds, or any components of the formulation
* Smoke more than 10 cigarettes or use the equivalent tobacco, smoking-cessation products, nicotine-containing products, or e cigarettes (nicotine and non nicotine) per day.
* Is a known user of drugs of abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2023-07-18 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Part A: Pharmacokinetics (PK): Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of LY3437943 | Predose on Day 1 up to 43 days postdose (Part A)
  Part A: PK: AUC(0-∞) of LY3437943
Part A: PK: Maximum Concentration (Cmax) of LY3437943 | Predose on Day 1 up to 43 days postdose (Part A)
  Part A: PK: Cmax of LY3437943

SECONDARY OUTCOMES:
Part B: PK: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of LY3437943 | Predose on Day 1 up to 71 days postdose (Part B)
  Part B: PK: AUC(0-∞) of LY3437943
Part B: PK: Maximum Concentration (Cmax) of LY3437943 | Predose on Day 1 up to 71 days postdose (Part B)
  Part B: PK: Cmax of LY3437943

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Fortrea Clinical Research Unit, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No